CLINICAL TRIAL: NCT05223452
Title: Role of Intestinal Ultrasound in Inflammatory Bowel Disease in Correlation to Endoscopic Findings
Brief Title: Role of Ultrasound in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shrouk Mohamed Gad, doctor, Assiut University
Other Study IDs: US IN IBD
Record Dates: First submitted 2021-10-23; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: UltraSound — we use prob that admit some of radiation to patient to see the organs inside the abdomen

SUMMARY:
The aim of this article is to provide an extensive overview of the actual role of bowel ultrasound in the detection and follow-up of patients with chronic inflammatory bowel disease

DETAILED DESCRIPTION:
The inflammatory bowel disease is a chronic bowel disorder; it can involve the whole gastrointestinal tract, but its localization in the ileum or colon is most common. The reference standard for the diagnosis of inflammatory bowel disease is ileocolonoscopy with histologic assessment. Dan Carter, Lior H. Katz, Eytan Bardan, Eti Salomon, Shulamit Goldstein, Shomron Ben Horin, Uri Kopylov, and Rami Eliakim The reference standard for the detection of any complications is surgery. However, imaging techniques have an important role both in the detection/localization of C D and in the followup of C D patients. In the last few years, the technical development of ultrasound equipment, the advent of new technologies such as elastography and mostly the increased expertise of sonographers have boosted the role of bowel ultrasound in assessment of the gastrointestinal tract. In fact, bowel ultrasound is particularly attractive thanks to its widespread availability, non-invasiveness, low cost and good reproducibility, as it can be easily repeated during follow-up Clara Benedetta Conti , Mariangela Giunta , Daniele Gridavilla , Dario Conte , Mirella Fraquelli . Bowel ultrasound has become the first-line imaging technique for patients with suspected C rohn's disease because it is cheap ,less radiation effect ,it can be done more than one time for follow up these patient . Some signs, for example, bowel loop elasticity (i.e., the capability of the bowel wall to collapse on the bowel lumen and return to the original size and shape after manual compression and decompression) and compressibility at probe contact and peristalsis (usually impaired), are not specific, whereas other signs, such as the characteristics of the bowel wall, are more specific. Among the latter, the most important sign is bowel wall thickening (BWT) . Also important are bowel wall echo pattern characteristics (BWP) , the presence of any margin irregularity and the grade of vascularity at echo color Doppler or power Doppler . Other yet less frequent signs are the luminal alterations, such as the distension or any luminal stenosis. Other possible findings outside the bowel loop are mesenteric hypertrophy , enlarged mesenteric lymph nodes and free fluid in the abdominal cavity or among the bowel loops .

ELIGIBILITY:
Inclusion Criteria:

* All patient reffered to radiology department for doing ultrasonography suspected to have bowel disease.

Exclusion Criteria:

* No patient excluded to do this process.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients that come to assuit university hospital suffering from bowel disease no exclusion
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
comparison of ultrasound findings with endoscopic findings | baseline
  analysis of ultrasound findings in patient and test if it can diagnose the different types of inflammatory bowel disease

REFERENCES:
- [Background] Andreoli A, Cerro P, Falasco G, Giglio LA, Prantera C. Role of ultrasonography in the diagnosis of postsurgical recurrence of Crohn's disease. Am J Gastroenterol. 1998 Jul;93(7):1117-21. doi: 10.1111/j.1572-0241.1998.00340.x. PMID 9672341
- [Background] Castiglione F, Bucci L, Pesce G, De Palma GD, Camera L, Cipolletta F, Testa A, Diaferia M, Rispo A. Oral contrast-enhanced sonography for the diagnosis and grading of postsurgical recurrence of Crohn's disease. Inflamm Bowel Dis. 2008 Sep;14(9):1240-5. doi: 10.1002/ibd.20469. PMID 18398896